CLINICAL TRIAL: NCT00828412
Title: A Randomized, Investigator-Blind, Six-Week, Parallel Group, Multicenter Pilot Study to Compare the Safety and Efficacy of EpiCeram Skin Barrier Emulsion and Desonide Cream 0.05% in the Twice Daily Treatment of Pediatric Subjects With Moderate Atopic Dermatitis
Brief Title: Comparison of the Efficacy and Safety of Two Topical Creams for Pediatric Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EPC0801
Record Dates: First submitted 2009-01-21; First posted 2009-01-26 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): EpiCeram Skin Barrier Emulsion
  Interventions: Device: EpiCeram Skin Barrier Emulsion
- 2 (Active Comparator): Desonide Cream 0.05%
  Interventions: Drug: Desonide Cream 0.05%

INTERVENTIONS:
Device: EpiCeram Skin Barrier Emulsion — topical cream, twice daily, 6 weeks
  Arms: 1
Drug: Desonide Cream 0.05% — topical cream, twice daily, 6 weeks
  Arms: 2

SUMMARY:
This study compares the effectiveness of two topical creams for atopic dermatitis in pediatric subjects. Subjects will be randomly assigned to use one of the two creams twice daily for 6 weeks or until clear.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 months of age and less than 13 years of age
* atopic dermatitis of moderate severity

Exclusion Criteria:

* pregnant or lactating
* treatment of atopic dermatitis with topical product in the 14 days prior to Baseline
* treatment of atopic dermatitis with systemic product in the 30 days prior to Baseline
* serious or uncontrolled medical condition
* active infection
* significant use of inhaled, intranasal, or intraocular corticosteroid

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Fraser, PhD, Study Director — Promius Pharma, LLC
Locations (5):
- United States (5):
  - National Jewish Health, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Dermatology Research Associates, Cincinnati, Ohio
  - University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- EpiCeram Skin Barrier Emulsion: EpiCeram Skin Barrier Emulsion topically twice daily
- Desonide Cream 0.05%: Desonide Cream 0.05% topically twice daily
Period: Overall Study
Arm/Group | EpiCeram Skin Barrier Emulsion | Desonide Cream 0.05%
Started | 50 | 50
Completed | 41 | 48
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Groups:
- EpiCeram Skin Barrier Emulsion: EpiCeram Skin Barrier Emulsion
- Desonide Cream 0.05%: Desonide Cream 0.05%
- Total: Total of all reporting groups
Arm/Group | EpiCeram Skin Barrier Emulsion | Desonide Cream 0.05% | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (3.5) | 4.8 (3.3) | 5.2 (3.4)
Gender [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 25 | 20 | 45
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100
Three item severity score [Mean (Standard Deviation); unit: units on a scale] — The average of the sum of scores for erythema, edema/papulation, and excoriation for two target lesions. Scoring on a scale of 0 to 3 (none to severe). Maximum score is 9.
  units on a scale | 5.4 (0.7) | 5.5 (0.7) | 5.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Three Item Severity Score
Description: The average of the sum of scores for erythema, edema/papulation, and excoriation for two target lesions. Scoring on a scale of 0 to 3 (none to severe). Maximum score is 9.
Time Frame: Baseline to 6 weeks
Population: All subjects with data were included in the analysis. No imputation was done for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EpiCeram Skin Barrier Emulsion: Week 6 EpiCeram Skin Barrier Emulsion
- Desonide Cream 0.05%: Week 6 Desonide Cream 0.05%
Arm/Group | EpiCeram Skin Barrier Emulsion | Desonide Cream 0.05%
Number analyzed (Participants) | 41 | 48
units on a scale | -2.6 (2.0) | -3.6 (1.8)

ADVERSE EVENTS:
Arm/Group | EpiCeram Skin Barrier Emulsion | Desonide Cream 0.05%
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 7/50 | 3/50
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EpiCeram Skin Barrier Emulsion (N=50) | Desonide Cream 0.05% (N=50)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Dernatitis atopic (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No